CLINICAL TRIAL: NCT04254601
Title: Red Low Level LASER Versus Narrow Band Ultraviolet B in the Treatment of Facial Acne Vulgaris
Brief Title: Laser Therapy Versus Narrow Band Ultraviolet B for the Treatment of Acne Vulgaris
Acronym: LLLT-NBUB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadaya Mosaad, Principal investigator., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/001693
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Skin Diseases
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Intervention Model Description: The present study is a pretest-post test single blind randomized controlled trial, conducted at Faculty of Physical Therapy, Cairo University.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental group 1 (Experimental): Patients in group (A) consisted of 15 participants, received a program of NBUB, DIXWELL EMLY 98 -ABRP 64 ,made in France (wavelength 311 to 313nm) , in addition to topical aknemycin medications (topical erythromycin cream 2% (Akne-Mycin- Egypt) two times per day on the entire face from the beginning to the end of the treatment period after 8 weeks).
  Interventions: Device: Narrow band ultraviolet B.; Drug: topical erythromycin cream 2% (Akne-Mycin- Egypt)
- Experimental group 2 (Experimental): Participants in-group (B) consisted of 15 participants, received a program of R-LLLT that was conducted through laser equipment InGaAs (630 nm, 10 mW, continuous) (RIKTA, Russia) with fluence 12 J/cm2, two sessions per week for 8 weeks Plus topical erythromycin cream 2% (Akne-Mycin- Egypt) two times per day on the entire face from the beginning to the end of the treatment period.
  Interventions: Device: Narrow band ultraviolet B.; Drug: topical erythromycin cream 2% (Akne-Mycin- Egypt)
- Control group (Active Comparator): Patients in the group C, consisted of 15 participants, were asked to apply topical erythromycin cream 2% (Akne-Mycin- Egypt) two times per day on the entire face from the beginning to the end of the treatment period.
  Interventions: Drug: topical erythromycin cream 2% (Akne-Mycin- Egypt)

INTERVENTIONS:
Device: Narrow band ultraviolet B. — NBUB: DIXWELL EMLY 98 -ABRP 64 ,made in France. Red LLL, InGaAs (630 nm, 10 mW, continuous) (RIKTA, Russia)
  Other Names: Red low level laser.
  Arms: Experimental group 1; Experimental group 2
Drug: topical erythromycin cream 2% (Akne-Mycin- Egypt) — two times per day on the entire face from the beginning to the end of the treatment period .
  The face is washed thoroughly with warm water and gentle soap, rinse well, and pat dry, patients were advised to wait 30 minutes before applying the aknemycin. To help keep new pimples from breaking out, the aknemycin was applied to the whole area usually affected by acne, not just to the pimples themselves

SUMMARY:
Forty-five participants with facial AV were assigned randomly to three groups of fifteen subjects each. Each group received various therapies. Group A (Study group A) had received both NBUB and akne-Mycin; Group B( study group B) had received Red LLLT and akne-Mycin and group C (Control group) received only akne-Mycin cream. All 45 participants are tested at the initial treatments, after 4 weeks and after 8 weeks by the acne count, the intensity scale and the photographic test.

DETAILED DESCRIPTION:
Forty-five patient (18 male and 27 female) were recruited on a referral basis from the department of dermatology at Kasr Al- aini Teaching Hospital. Firstly, an interview was held with each participant to determine gender, age, skin type, acne severity and medical prescriptions,Randomization was performed by selecting numbers from opaque envelopes containing numbers that were chosen by a random number generator, selection was done by an independent person.

Patients in group (A) received a program of NBUB, ( DIXWELL EMLY 98 -ABRP 64 ,made in France) wavelength 311 to 313nm , in addition to topical aknemycin medications. Each treatment lasts one to eight minutes. The treatments were given three times a week. for 8 weeks.Participants in-group (B) received a program of R-LLLT that was conducted through laser equipment InGaAs (630 nm, 10 mW, continuous) (RIKTA, Russia) with fluence 12 J/cm2, two sessions per week for 8 weeks .Patients in the three groups were asked to apply topical erythromycin cream 2% (Akne-Mycin- Egypt) two times per day on the entire face from the beginning to the end of the treatment period .Evaluation was based on formal counts of active lesions (papule and pustule).facial photographs using a digital camera (PANASONIC, Tokyo, Japan). and Five-point scale of investigators assessment that reflect lesion count improved percentage.

ELIGIBILITY:
Inclusion Criteria:

* Ages ranged from 18-35 years.
* Skin type III and IV.
* Mild to moderate facial acne.

Exclusion Criteria:

* Treatment with oral retinoid within past 1 year.
* Treatment with other acne treatment within past 3 months.
* History of treatment with systemic and topical antibiotics for acne vulgaris within the last 1 month.
* Treatment with oral isotretinoin within the last 6 months.
* Participants received radiotherapy or chemotherapy.
* Any history of photosensitivity.
* Chemical peels during the previous 4 weeks.
* Seizures,
* Pregnancy
* Use of oral contraceptives.
* Breastfeeding .

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
formal counts of active acne lesions. | 8 weeks.
  The lesion number was individually counted by lesion type at all three times of evaluation as the number of papules and pustules

SECONDARY OUTCOMES:
facial photographic method. | 8 weeks.
  facial photographs using a digital camera (PANASONIC, Tokyo, Japan). Photos of the front and bilateral sides of the face were clinically taken each time, by same manner at all time points.

OTHER OUTCOMES:
lesion count changed percentage. | 8 weeks.
  Five-point scale of investigators assessment that reflect lesion count changed percentage; worse: < - 10 percent, no change:_9percent-9percent, mild improvement: 10percent-39percent, moderate improvement: 40percent-59percent, marked improvement: 60percent-89percent, and clearance: ≥-90percent.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP
Time Frame: we will share the study after 6 months of publication.

REFERENCES:
- [Derived] Eid MM, Saleh MS, Allam NM, Elsherbini DM, Abdelbasset WK, Eladl HM. Narrow Band Ultraviolet B Versus Red Light-Emitting Diodes in the Treatment of Facial Acne Vulgaris: A Randomized Controlled Trial. Photobiomodul Photomed Laser Surg. 2021 Jun;39(6):418-424. doi: 10.1089/photob.2020.4988. Epub 2021 May 20. PMID 34015228